CLINICAL TRIAL: NCT05578963
Title: Corelation Between Palmaris Longus Muscle and Carpel Tunnel Syndrome in Health Profession Students Across Pakistan
Brief Title: Correlation Between Palmaris Longus Muscle and Carpel Tunnel Syndrome
Status: Completed | Type: Observational
Sponsor: Bahria University (Other)
Responsible Party: Principal Investigator, Seyyada Tahniat Ali, clinical instructor, Bahria University
Other Study IDs: FRC-BUMDC35/2021
Record Dates: First submitted 2022-10-11; First posted 2022-10-13 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Schaeffer's Test for palmaris tendon — After demographics, Schaeffer's Test will be used to check the presence or absence of palmaris longus muscle. In this test, students will maintain the forearm at 90 degrees first followed by moving the thumb in opposition towards the little finger with the wrist partially flexed. If the tendon bulges out, it will reflect presence of palmaris longus and vice versa. This finding will be recorded. After that, students will perform Phalen's test. In this test, researcher will ask them to press the backs of their hands and fingers together with their wrists flexed and fingers pointed down. they'll stay that way for a minute or two. If fingers tingle or get numb, it will indicate carpal tunnel syndrome. The reading will be recorded.
  Other Names: Phalen test for carpel tunnel syndrome

SUMMARY:
The Palmaris longus (PL) muscle is a long, adaptable muscle that lies between the Flexor Carpi Ulnaris and Flexor Carpi Radialis muscles in the shallow volar segment of the lower arm. It has been acknowledged as a minimal muscle, nonetheless, in light of the fact that reviews have uncovered that around 30% of the populace might be feeling the loss of this muscle in one lower arm (one-sided) or the two lower arms (reciprocal), but the rate could continuously fluctuate. Carpal tunnel syndrome is an often-observed disease that causes pain, numbness, and tingling in the hand and arm. The disease occurs when one of the major nerves to the hand - the median nerve - is compressed as it moves across the wrist. The abnormal passage of palmaris longus tendon through the carpal tunnel leads to a contributory factor for causing the median nerve compression.

DETAILED DESCRIPTION:
The Palmaris longus (PL) muscle is a long, adaptable muscle that lies between the Flexor Carpi Ulnaris and Flexor Carpi Radialis muscles in the shallow volar segment of the lower arm. It has been acknowledged as a minimal muscle, nonetheless, in light of the fact that reviews have uncovered that around 30% of the populace might be feeling the loss of this muscle in one lower arm (one-sided) or the two lower arms (reciprocal), but the rate could continuously fluctuate. Agenesis is a typical physical variety. Hold strength is unaffected by the deficiency of the palmaris longus. Past examination has assessed that 15% of the worldwide populace has palmaris longus ligament agenesis (PLA), which is more successive in ladies and has an affinity to be higher respectively however, if present singularly, is normally on the left side. It emerges from the Medial Epicondyle of the Humerus and goes into the Palmar Aponeurosis and Flexor Retinaculum at the wrist joint through the normal flexor ligament. It accepts its innervation from the Median Nerve. Palmaris longus works couple with the lower arm's long flexors to give flexion at the wrist joint and small joints of the hand. The muscle additionally helps in fixing and worrying the palmar aponeurosis.

Carpal tunnel syndrome is an often-observed disease that causes pain, numbness, and tingling in the hand and arm. The disease occurs when one of the major nerves to the hand - the median nerve - is compressed as it moves across the wrist. The abnormal passage of palmaris longus tendon through the carpal tunnel leads to a contributory factor for causing the median nerve compression. The tendinous structure normally passes anterior to the flexor retinaculum and then distally continues with the palmar aponeurosis. This topographic relationship of the tendon with the median nerve makes its anatomical variations a common cause of median nerve entrapment. Several anatomical variations of the PL muscle have been studied in the past. The variations could be in the form of complete absence, insertion site variation, multiple muscle bellies, different location of the muscle belly, and so on.

ELIGIBILITY:
Inclusion Criteria:

* Health profession Students with carpel tunnel syndrome across Pakistan
* Age should be 18-23 years

Exclusion Criteria:

* Students who had carpel tunnel release surgery
* Any wrist related pathology
* Involve in any other wrist related research
* Underwent any surgery of wrist
* Underwent any surgery that required replacement of tendon
* Underwent any surgery that had Palmaris longus tendon for replacement

Ages: 18 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: • Health profession Students with carpel tunnel syndrome across Pakistan
Sampling Method: Non-Probability Sample
Enrollment: 258 (Actual)
Dates: Start 2022-10-15 (Actual); Primary Completion 2024-11-25 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
correlation of palmaris longus tendon and carpel tunnel syndrome | 1 day
  The first test developed in 1909. It Involves maintaining the forearm at 90 degrees first followed by moving the thumb in opposition towards the little finger with the wrist partially flexed. The building tendon represents the presence of palmaris longus muscle.The practitioner will tell you to press the backs of your hands and fingers together with your wrists flexed and your fingers pointed down. You'll stay that way for a minute or two. If fingers tingle or get numb, it indicates carpal tunnel syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Seyyada T Ali, Principal Investigator — Bahria university health sciences campus
Locations (1):
- Seyyada Tahniat Ali, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clinical Assessment of the Palmaris Longus - Accuracy of common tests Authors: Kigera JWM1 MBChB, MMed (Ortho), Mukwaya S2 Affiliation
- [Background] Priganc VW, Henry SM. The relationship among five common carpal tunnel syndrome tests and the severity of carpal tunnel syndrome. J Hand Ther. 2003 Jul-Sep;16(3):225-36. doi: 10.1016/s0894-1130(03)00038-3. PMID 12943125
- [Result] Mohammad WS. Work-related risk factors for Carpal Tunnel Syndrome among Majmaah University female touchscreen users. Pak J Med Sci. 2019 Sep-Oct;35(5):1221-1226. doi: 10.12669/pjms.35.5.683. PMID 31488982